CLINICAL TRIAL: NCT03916536
Title: Holmium Laser Versus Thulium Laser Versus Bipolar Enucleation of the Prostate for Treatment of Large Sized Benign Prostatic Enlargement. A Randomized Controlled Trial
Brief Title: Holmium Laser Versus Thulium Laser Versus Bipolar Enucleation of the Prostate.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Fady kamal Ghobrial, principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prostate Enucleation
Record Dates: First submitted 2019-04-13; First posted 2019-04-16 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Prostate Hypertrophy; Holmium Laser; Thulium Laser; Bipolar Diathermy; Prostate Enucleation
Keywords: Holmium Laser; Thulium Laser; Bipolar diathermy; prostate enucleation
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Holmium Laser (Active Comparator): holmium laser enucleation of the prosteate
  Interventions: Procedure: Holmium Laser
- Thulium Laser (Active Comparator): Thulium laser enucleation of the prosteate
  Interventions: Procedure: Thulium Laser
- Bipolar Enucleation (Active Comparator): Bipolar enucleation of the prosteate
  Interventions: Procedure: Bipolar diathermy

INTERVENTIONS:
Procedure: Holmium Laser — Holmium laser enucleation of large sized prostate
  Other Names: HoLEP
  Arms: Holmium Laser
Procedure: Thulium Laser — Thulium laser enucleation of large sized prostate
  Other Names: ThuLEP
  Arms: Thulium Laser
Procedure: Bipolar diathermy — Bipolar enucleation of large sized prostate
  Other Names: Bipolar enucleation
  Arms: Bipolar Enucleation

SUMMARY:
Because of the diversity of the studies and deficiency of those comparing various techniques of EEP for treatment of LUTs secondary to BPO in patients with large sized prostate, we aim in this study at testing the non-inferiority of PKEP and ThuLEP to HoLEP in relieving LUTs secondary to BPO in patients prostate size >80ml. Our hypothesis is to present an evidence that enucleation is a technique rather than a power dependent procedure through a RCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age >50 years
* Lower urinary tract symptoms LUTS secondary benigh prostatic obstruction BPO who failed medical treatment
* International prostate symptom scores (IPSS) >15 and bother score quality of life (QOL) > 3 (according to IPSS question 8)
* Maximum urinary flow rate (Q max) <15 ml/sec with at least 150 ml voided volume or cases with acute urine retention secondary to BPO who failed trial of voiding on medical treatment.
* Transrectal ultrasound TRUS estimated total prostate size 80-250cc

Exclusion Criteria:

* Patient with neurological disorder which might affect bladder function as cerebrovascular stroke, Parkinson disease
* Active urinary tract infection (positive urine culture) till treatment
* Presence of bladder cancer (within the last 2 years)
* Known prostate cancer patients will be excluded preoperatively on the basis of digital rectal examination, prostate specific antigen level, and TRUS imaging followed by prostate biopsies if necessary.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 155 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
urinary functional outcomes using uroflowmetry | 2 years
  assessed by maximum flow rate (Q-max) measured using uroflowmetry by ml/sec, better outcome above 15ml/sec

SECONDARY OUTCOMES:
patient symptoms | 2 years
  assessed by international prostate symptoms score (IPSS) questionnaire, better outcome score below 9
perioperative complications | 2 years
  assessed by clavien dindo score

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shoma AM, Ghobrial FK, El-Tabey N, El-Hefnawy AS, El-Kappany HA. A randomized trial of holmium laser vs thulium laser vs bipolar enucleation of large prostate glands. BJU Int. 2023 Dec;132(6):686-695. doi: 10.1111/bju.16174. Epub 2023 Sep 28. PMID 37667842